CLINICAL TRIAL: NCT05176821
Title: Eradication Efficacy and Safety of High-dose Dual Therapy Compared With Furazolidone-based Quadruple Therapy as a Rescue Treatment for Helicobacter Pylori Infection: a Randomized Controlled Trial
Brief Title: Eradication Efficacy and Safety of Two Rescue Treatments for Helicobacter Pylori Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JW-Hp2021
Record Dates: First submitted 2021-12-14; First posted 2022-01-04 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: H. Pylori Infection
MeSH Terms: interventions — Esomeprazole; Amoxicillin; Furazolidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-dose dual therapy group (Experimental): esomeprazole 20mg qid plus amoxicillin 750mg qid were used in the high-dose dual therapy group
  Interventions: Drug: esomeprazole plus amoxicillin
- Furazolidone-based quadruple therapy (Active Comparator): furazolidone 100mg bid + amoxicillin 1000mg bid + esomeprazole 20mg bid + bismuth potassium citrate 1000mg(220mg of bismuth) bid were used in the Furazolidone-based quadruple therapy
  Interventions: Drug: amoxicillin, furazolidone, bismuth potassium citrate , esomeprazole

INTERVENTIONS:
Drug: esomeprazole plus amoxicillin — amoxicillin 750mg QID + esomeprazole 20mg QID for 14 days
  Other Names: HDDT
  Arms: High-dose dual therapy group
Drug: amoxicillin, furazolidone, bismuth potassium citrate , esomeprazole — amoxicillin 1000mg BID + furazolidone 100mg BID + bismuth potassium citrate 600mg BID + esomeprazole 20mg BID for 14 days
  Other Names: FT
  Arms: Furazolidone-based quadruple therapy

SUMMARY:
The aim of this study was to evaluate the efficacy and safety of high-dose dual therapy compared with furazolidone-based quadruple therapy as a rescue treatment for helicobacter pylori infection.

DETAILED DESCRIPTION:
Helicobacter pylori (H. pylori) infection is common worldwide and is strongly associated with peptic ulcer and gastric cancer. The eradication rate of H. pylori treatment is limited in the recent years although standard first-line therapy is used. There is a growing antibiotic resistance due to antibiotic consumption for other infections. The failure of first-line therapy for H. pylori can significantly limit the efficacy of the subsequent rescue therapies.

H. pylori resistance to amoxicillin (AMO), both primary and acquired, have been reported to be uncommon. The bactericidal effect of AMO against H. pylori is pH- and time- dependent with a sustaining higher intragastric pH. Thus, the therapy consisting of high-dose PPI and AMO may have advantage over the currently recommended furazolidone-based quadruple therapy.

ELIGIBILITY:
Inclusion Criteria:

* The patients who were diagnosed with persistent H. pylori infection and had previously failed one or more courses of eradication therapies that included amoxicillin, clarithromycin, or nitroimidazole.

Exclusion Criteria:

* Age < 18 years old.
* The time frame was less than 6 months from the previous eradication therapy.
* The previous eradication therapy included furazolidone.
* Allergic to the medication.
* Pregnant or lactating women.
* Comorbidities of severe conditions like hepatic, renal or cardiorespiratory diseases or malignancy.
* Administration of antibiotics, bismuth or PPI in the preceding 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
eradication rate | 42 days
  eradication rate of H pylori, presenting with negative results on the 13C-UBT test

SECONDARY OUTCOMES:
frequency of the adverse events | 42 days
  incidence rate of the adverse events, including dyspepsia, nausea, vomiting, abdominal pain, bloating, diarrhea, dizziness, headache, skin rash, fatigue and fever.
compliance rate of the drugs | 42 days
  Compliance was defined as good when they had taken more than 80% of the total medication.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Jiang, MD, Principal Investigator — Xiamen branch of Zhongshan Hospital, Fudan University
Locations (1):
- Zhongshan Hospital Xiamen Branch, Xiamen, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available to other researchers. We may balance the potential benefits and risks for each request and then provide the data that could be shared.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available once the results have been uploaded in the PRS system and will be available for 2 years.
Access Criteria: Emails could be sent to the emails below to obtain the shared data: chen.jie5@zs-hospital.sh.cn, weng.chengzhao@zsxmhospital.com

REFERENCES:
- [Background] Yang J, Zhang Y, Fan L, Zhu YJ, Wang TY, Wang XW, Chen DF, Lan CH. Eradication Efficacy of Modified Dual Therapy Compared with Bismuth-Containing Quadruple Therapy as a First-Line Treatment of Helicobacter pylori. Am J Gastroenterol. 2019 Mar;114(3):437-445. doi: 10.14309/ajg.0000000000000132. PMID 30807294
- [Background] Yu L, Luo L, Long X, Liang X, Ji Y, Graham DY, Lu H. High-dose PPI-amoxicillin dual therapy with or without bismuth for first-line Helicobacter pylori therapy: A randomized trial. Helicobacter. 2019 Aug;24(4):e12596. doi: 10.1111/hel.12596. Epub 2019 May 20. PMID 31111580